CLINICAL TRIAL: NCT02812979
Title: Evaluation of the Effectiveness of the Nebulization Bronchodilators Under High Nasal Flow Humidified Compared to a Usual Method
Brief Title: Evaluation of the Effectiveness of the Nebulization Bronchodilators Under High Nasal Flow Humidified
Acronym: AirvoNEB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PHAO15-SE / AirvoNEB; 2016-A00064-47 (Other: ID RCB)
Record Dates: First submitted 2016-06-16; First posted 2016-06-24 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2018-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Masks

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Airvo2 with Aerogen Solo (Experimental): AIRVOTM2 will be set to deliver air (21% oxygen concentration ) at a rate of 30 L / min at 100 % relative humidity at 37 ° C.
  Nebulization of salbutamol will be effected by means of a nebulizer to the vibrating screen (Aerogen® Solo, Aerogen , Galway, Ireland ) which is a nebulizing device for single use, commonly used in invasive and non invasive mechanical ventilation.
  Nebulizer will be responsible for a salbutamol solution available in the form of containers of 2.5 ml containing 2.5 mg of salbutamol
  Interventions: Device: Airvo2 with Aerogen Solo
- Mask (Active Comparator): During nebulization in the usual way ( oral facial mask ) , it will be used a pneumatic nebulizer powered by a 6 L / min air flow rate ( usual method ).
  Nebulizer will be responsible for a salbutamol solution available in the form of containers of 2.5 ml containing 2.5 mg of salbutamol
  Interventions: Device: Mask
- arm control Airvo2 without nebulization of salbutamol (Placebo Comparator): control procedure is to be placed under humidified high flow nasal alone
  Interventions: Device: arm control Airvo2 without nebulization of salbutamol

INTERVENTIONS:
Device: Airvo2 with Aerogen Solo — Nebulization of salbutamol with Airvo 2 and Aerogen solo
  Other Names: AirvoNEB
  Arms: Airvo2 with Aerogen Solo
Device: Mask — Usual nebulization of salbutamol with mask
  Arms: Mask
Device: arm control Airvo2 without nebulization of salbutamol — Airvo2 with Aerogen Solo. No nebulization of salbutamol
  Arms: arm control Airvo2 without nebulization of salbutamol

SUMMARY:
The principal objective is to show noninferiority of nebulized salbutamol through the high flow nasal system moistened AIRVO ™ 2 in terms of reversibility of airflow obstruction compared to nebulization by the usual method (spray mask).

DETAILED DESCRIPTION:
Randomized, comparative, non inferiority study between two nebulization strategies bronchodilators, one according to the method tested namely the spray - in across the top humidified nasal flow system and the other according to a customary procedure, through a mask. A third arm will be evaluated (control arm) to overcome a possible own bronchodilator effect of high flow nasal humidified.

ELIGIBILITY:
Inclusion Criteria:

* adults
* Patient with chronic obstructive pulmonary disease
* Patients, when performing lung function tests performed outside of the study :

  1. A report FEV / FVC less than 60% prior to bronchodilator treatment AND
  2. A positive reversal test defined by FEV variation of over 12 % and 200 mL after administration of inhaled salbutamol
* Patients affiliated to social security scheme
* Informed consent signed by the patient

Exclusion Criteria:

* Exacerbation of chronic obstructive pulmonary disease during
* Uncontrolled asthma
* Pneumothorax current or recent ( < 2 months)
* Pleural aspiration or biopsy , trans - bronchial biopsies and / or bronchoalveolar lavage in the preceding 48h
* hemoptysis in progress
* Patient under guardianship or trusteeship safeguard justice
* Pregnant or breastfeeding women or parturient woman
* Known allergy or intolerance to salbutamol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-06; Primary Completion 2018-04-27 (Actual); Study Completion 2018-04-27 (Actual)

PRIMARY OUTCOMES:
Increased expiratory volume in one second ( FEV ) | measured before and after nebulization of salbutamol at 0 minute and 15 minutes after nebulization of salbutamol

SECONDARY OUTCOMES:
clinical data (FVC) on the physiological effects of high nasal flow | before and after treatment with humidified high nasal flow at 0 minute and 30 minutes after the treatment with humidified high nasal flow
clinical data (FEV) on the physiological effects of high nasal flow | before and after treatment with humidified high nasal flow at 0 minute and 30 minutes after the treatment with humidified high nasal flow
clinical data (FEV / FVC) on the physiological effects of high nasal flow | before and after treatment with humidified high nasal flow at 0 minute and 30 minutes after the treatment with humidified high nasal flow

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Réanimation Polyvalente, Tours, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Reminiac F, Vecellio L, Bodet-Contentin L, Gissot V, Le Pennec D, Salmon Gandonniere C, Cabrera M, Dequin PF, Plantier L, Ehrmann S. Nasal high-flow bronchodilator nebulization: a randomized cross-over study. Ann Intensive Care. 2018 Dec 20;8(1):128. doi: 10.1186/s13613-018-0473-8. PMID 30570679